CLINICAL TRIAL: NCT06315556
Title: Drug Utilization Study for Eylea 40 mg/mL Using the PICLEO Paediatric Dosing Device in Preterm Infants With Retinopathy of Prematurity in the UK
Brief Title: An Observational Study to Collect Data on How Aflibercept (Eylea) Given Using a Paediatric Dosing Device is Used in Preterm Babies With Retinopathy of Prematurity in the United Kingdom (UK)
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22539
Record Dates: First submitted 2024-02-26; First posted 2024-03-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Retinopathy of Prematurity; Preterm Infants
Keywords: ROP
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature infants diagnosed with ROP: Premature infants diagnosed with retinopathy of prematurity (ROP) and treated with aflibercept 0.4 mg using the Eylea 40 mg/mL prefilled syringe (PFS) in combination with the PICLEO paediatric dosing device (PDD) after marketing authorisation in UK and included in the National Neonatal Research Database (NNRD).
  Interventions: Drug: Aflibercept (Eylea)

INTERVENTIONS:
Drug: Aflibercept (Eylea) — Eylea 40 mg/mL solution for injection in pre-filled syringe.

SUMMARY:
This is an observational study in which only data from babies with retinopathy of prematurity (ROP) who are being treated with aflibercept (Eylea) in prefilled syringe (PFS) using a paediatric dosing device (PDD) are collected and studied.

ROP is a condition that affects the eyes of preterm babies. It occurs when the baby's retina, the part of the eye that senses light, does not develop normally. This may result in vision problems, including blindness, if left untreated. Preterm babies are born before 37 weeks of pregnancy. ROP is more likely to develop in babies who are born before 32 weeks of pregnancy or weigh less than 1.5 kilograms at birth.

Aflibercept is a drug that is injected into the eye. It works by blocking a protein called vascular endothelial growth factor (VEGF) which causes abnormal growth of blood vessels in the retina.

Aflibercept in PFS given using a PDD is approved for the treatment of babies with ROP. The prefilled syringe will be fitted with an injection needle to give aflibercept. And a PDD is a tool used to give the right amount of aflibercept to children in a safe manner.

Since there are other treatments which are commonly used for babies with ROP, the extent of use of aflibercept given using a PDD is unknown.

The main purpose of this study is to:

* find the number of preterm babies who are treated with aflibercept using a PDD in the UK
* inform whether this number is enough to perform a study to learn about the long-term safety of aflibercept given using a PDD in babies with ROP

An additional purpose of this study is to describe characteristics including age, sex, and race, and signs and symptoms of ROP observed in babies being treated with aflibercept using a PDD.

The data will come from a database called the National Neonatal Research Database. The study will cover the period from March 2024 to March 2025, if the number of babies found is enough to perform the safety study. If not, data will be collected till April 2027.

In this study only available data from preterm babies born during the study period are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible infants within the NNRD include those who were:

  * 1. Born during the study period, i.e. from Q4/2023 following market introduction of Eylea PFS+PDD and 31st December 2026, and
  * 2. Received care in a neonatal unit that contributes data to the NNRD and the unit has agreed to participate in the study, and
  * 3. Diagnosed with ROP in any stage in at least one eye.

Exclusion Criteria:

* Infants with missing data for gestational age at birth will be excluded.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All premature infants diagnosed with ROP and treated with Eylea PFS + PDD included in the National Neonatal Research Database (NNRD) during the study period in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated with Eylea PFS+PDD upon completion of 1- or 3-years following market introduction | From market introduction of Eylea PFS+PDD in UK up to 3 years
  * To evaluate trends in drug utilization patterns of Eylea prefilled syringe (PFS)+Paediatric Dosing Device (PDD) in the ROP patient population. Exposure to Eylea is defined as a record of Eylea PFS+PDD in the National Neonatal Research Database (NNRD) database during admission to the neonatal unity during the study period.
  * To inform the decision on whether the number of preterm infants with ROP exposed to Eylea PFS+PDD is sufficient (n=200) for proceeding with a cohort study to collect data on long-term safety (ocular and systemic safety including neurodevelopmental outcome).

SECONDARY OUTCOMES:
Summary of patient characteristics reported as number of participants with different categories | From market introduction of Eylea PFS+PDD in UK up to 3 years
  Birth weight (in categories), sex, gestational age in weeks (in categories), ethnicity, etc.
Summary of maternal factors reported as number of participants with different categories | From market introduction of Eylea PFS+PDD in UK up to 3 years
  Problems during pregnancy with mother, problems during pregnancy, mode of delivery, meconium stained liquor at delivery, etc.
Summary of comorbidities reported as number of participants with different categories | From market introduction of Eylea PFS+PDD in UK up to 3 years
  Brain injury, necrotising enterocholitis, pulmonary hemorrhage, chronic lung disease, etc.
Summary of clinical condition and resource utilization reported as number of participants with different categories | From market introduction of Eylea PFS+PDD in UK up to 3 years
  Respiratory support (mode of ventilation), cardiovascular (inotropic support), feeding (parenteral and enteral nutrition)
Summary of clinical condition and resource utilization reported as days | From market introduction of Eylea PFS+PDD in UK up to 3 years
  Intensive care days, invasive ventilation days, parenteral nutrition days
Summary of outcomes of the premature infants reported as number of participants with different categories | From market introduction of Eylea PFS+PDD in UK up to 3 years
  Survival to discharge from neonatal care (Y/N); Discharge, death, transferred to another hospital (in categories)
Summary of ocular disease and treatment reported as number of participants with different categories | From market introduction of Eylea PFS+PDD in UK up to 3 years
  Number of Eylea injections in the neonatal unity, ROP surgery, ROP stage, ROP clock hours, ROP Max zone, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.